CLINICAL TRIAL: NCT00105794
Title: Psychiatric Advance Directives for Improved Healthcare
Brief Title: Psychiatric Advance Directives for Improved Mental Health Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: PCC 02-054
Record Dates: First submitted 2005-03-16; First posted 2005-03-17 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2007-06

CONDITIONS: Schizophrenia; Schizoaffective; Bipolar Disorder; Stress Disorders, Post-traumatic; Psychotic Disorders
Keywords: advance directives; advance directive adherence; patient-centered care; patient satisfaction; coercion; informed consent; commitment of mentally ill; physician-patient relations
MeSH Terms: conditions — Schizophrenia; Bipolar Disorder; Stress Disorders, Post-Traumatic; Psychotic Disorders; Patient Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Other)
  Interventions: Procedure: Psychiatric Advance Directives intervention

INTERVENTIONS:
Procedure: Psychiatric Advance Directives intervention

SUMMARY:
During a psychiatric crisis, persons with severe mental illness (SMI) confront complex challenges concerning treatment choices and are often ill equipped or unable to make mental health care decisions. Psychiatric Advance Directives (PADs) are legal documents that allow competent persons to declare their treatment preferences in advance of a mental health crisis, when they may lose capacity to make reliable health care decisions. The use of PADs is consistent with recommendations of the President�s New Freedom Commission on Mental Illness and the Patient Self-Determination Act; 25 states have now adopted PAD legislation. VA does not have a specific policy for PADs or mechanisms to notify veterans of their right to prepare PADs. The downstream effects of PADs on patient care, crisis management, service use, and clinical outcomes are unknown.

DETAILED DESCRIPTION:
Background:

During a psychiatric crisis, persons with severe mental illness (SMI) confront complex challenges concerning treatment choices and are often ill equipped or unable to make mental health care decisions. Psychiatric Advance Directives (PADs) are legal documents that allow competent persons to declare their treatment preferences in advance of a mental health crisis, when they may lose capacity to make reliable health care decisions. The use of PADs is consistent with recommendations of the President�s New Freedom Commission on Mental Illness and the Patient Self-Determination Act; 25 states have now adopted PAD legislation. VA does not have a specific policy for PADs or mechanisms to notify veterans of their right to prepare PADs. The downstream effects of PADs on patient care, crisis management, service use, and clinical outcomes are unknown.

Objectives:

This project examined the effects of a facilitated PAD intervention on guiding patients� treatment during a future mental health crisis, patients� treatment engagement, and patients� mental health service use and clinical outcomes. An additional objective was to describe veterans� preferences for PAD content and completion. Study hypotheses predicted that, as compared to controls, veterans with PAD would have fewer involuntary hospitalizations, great satisfaction with care, less coercion and more autonomy, greater treatment motivation, stronger working alliances, less ER use and fewer rehospitalizations, and improved clinical outcomes.

Methods:

A total of 240 psychiatrically hospitalized veterans with severe mental illness were enrolled in this prospective, randomized, clinical intervention trial: 120 were randomized to �usual care� and received information about PADs; 120 were randomized to the PAD condition. All participants and their clinicians received information about PADs. Those randomized to the PAD condition were also offered the opportunity to complete a facilitated PAD. The facilitated PAD consisted of a 60-minute meeting with a clinician, who provided education about PADs and conducted a semi-structured interview to assess the patient�s wishes and preferences for future treatment during a mental health crisis. The clinician then assisted the patient to prepare a PAD document. Patients in both groups completed follow-up assessments at 1, 6, and 12 months post-enrollment. Those rehospitalized at Durham VAMC during the 12-month follow up period completed an additional assessment interview at each rehospitalization.

Status:

Complete. Activities completed in the past 12 months include collection of follow-up data on final subset of enrollees, extraction of utilization data (clinic stops) at one-year post-enrollment from VA system healthcare database (Austin, TX) and from local healthcare database (CPRS), completion of statistical analyses of outcome measures and preparation of scientific reports summarizing final results.

ELIGIBILITY:
Inclusion Criteria:

veteran diagnosis of schizophrenia, schizoaffective disorder, psychosis NOS, major depression with psychosis, bipolar I, PTSD.

At enrollment, hospitalized at the Durham VAMC psychiatric inpatient unit and receiving or anticipating outpatient treatment at the Durham or Raleigh VA facilities after discharge.

Exclusion Criteria:

Not competent (dementia, guardian, does not pass competency screen) Not followed in VA system for mental health care or available for follow-uo.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2004-03; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Rate of involuntary commitment (12 months), perceived coercion (baseline, 1, 6, 12, and rehospitalization), and treatment adherence (baseline and 12 months and record review)

SECONDARY OUTCOMES:
Satisfaction with inpatient care (baseline, rehospitalization), treatment motivation, working alliance, psychiatric symptoms, PAD completion, PAD content, PAD consulted (hospital record review), psychiatric ER use (12 month record review).

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer L. Strauss, BA MS PhD, Principal Investigator — Durham VA Medical Center, Durham, NC
Locations (1):
- Durham VA Medical Center, Durham, NC, Durham, North Carolina, United States

REFERENCES:
- [Result] Zervakis JB, Stechuchak KM, Olsen MK, Swanson JW, Oddone EZ, Weinberger M, Bryce ER, Butterfield ML, Swartz MS, Strauss JL. Previous Involuntary Commitment is Associated with Current Perceptions of Coercion in Voluntarily Hospitalized Patients. International Journal of Forensic Mental Health. 2007 Nov 1; 6(No. 2):105-112.
- See also: Click here for more information about this study: Psychiatric Advance Directives for Improved Healthcare — http://www.hsrd.research.va.gov/research/abstracts.cfm?Project_ID=2141692550&UnderReview-no